CLINICAL TRIAL: NCT02257645
Title: A Multicenter, Post-authorization Safety Study of Euforvac-Hib Vaccine for Active Primary Immunization Against Diphtheria, Tetanus, Pertussis, Hepatitis B and Haemophilus Influenza Type B in Infants
Brief Title: Post-authorization Safety Study of Euforvac-Hib Vaccine for Active Primary Immunization in Infants From 6 Weeks
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: LG Life Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: LG-VFOS001
Record Dates: First submitted 2014-10-02; First posted 2014-10-06 (Estimated); Last update posted 2014-10-07 (Estimated); Status verified 2014-10

CONDITIONS: Diphtheria; Tetanus; Pertussis; Hepatitis B; Haemophilus Influenza Type B
MeSH Terms: conditions — Diphtheria; Tetanus; Whooping Cough; Hepatitis B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Euforvac-Hib vaccine

SUMMARY:
A multicenter, observational study to evaluate the safety of Euforvac-Hib vaccine for active primary immunization against diphtheria, tetanus, pertussis, hepatitis B and Haemophilus influenza type B in infants.

DETAILED DESCRIPTION:
Euforvac-Hib vaccine manufactured by LG Life science in Korea, but it's not marketed in Korea. It is distributed to UN agencies in diverse countries. Thus, WHO recommended LG Life Science to conduct the safety study for assessing the vaccine safety if Euforvac-Hib is prequalified.

The objectives of this safety study are to identify any problems and questionable issues likely to emerge from the actual use of Euforvac-Hib vaccine after launching in the market.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who had been signed informed consent by subjects legally acceptable Representative
2. Infant from 6 weeks of age.who is given this vaccine for active primary immunization against diphtheria, tetanus, pertussis, hepatitis B and Haemophilus influenza type B

Exclusion Criteria:

1. Patients with hypersensitivity to any component for the vaccine
2. Patients who had a severe reaction to a previous dose of the combination vaccine or any of its constituents is absolute contraindication to subsequent doses of the combination vaccine.
3. Patients who had pertussis, encephalopathy or other serious neurological abnormality in the newborn period

Min Age: 6 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Infant from 6 weeks of age.who is given this vaccine for active primary immunization against diphtheria, tetanus, pertussis, hepatitis B and Haemophilus influenza type B
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-05 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Adverse event | up to 12 weeks after vaccination